CLINICAL TRIAL: NCT06174077
Title: Interest of Continuous Monitoring of the Fluoroscopy Time on the Dose Delivered to the Patient During Vertebral Cementoplasty Gestures With a Flat Panel Detector
Brief Title: Monitoring of Fluoroscopy Time on the Dose Delivered to the Patient During Vertebral Cementoplasty Procedures
Acronym: CIMVER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7993
Record Dates: First submitted 2022-11-29; First posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Vertebra Compression Fracture
Keywords: Vertebra Compression Fracture; Vertebral cementoplasty; Fluoroscopy time; Fluoroscopic control; Single-level vertebral cementoplasty

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The interventional radiology department of the Strasbourg University Hospital performs approximately 1,000 vertebral cementoplasties per year. This is one of the most practiced procedures in the department and therefore exposes the professionals in the room to significant annual cumulative doses of irradiation.

The objective of the study is to evaluate the interest of continuous visual monitoring of the fluoroscopy time by the operator on the dose delivered to the patient during an interventional radiology procedure performed under fluoroscopic control. The chosen reference examination is a single-level vertebral cementoplasty, a standardized examination that is frequent enough to allow easy data collection

ELIGIBILITY:
Inclusion criteria:

* Adult patient (≥18 years old)
* Man or woman
* Patient cared for at the HUS in interventional service for the realization of a vertebral cementoplasty of a single level between 01/06/2020 and 30/09/2020
* Subject who has not expressed his opposition, after being informed, to the reuse of his data for the purposes of this research.

Exclusion criteria:

* Patient who expressed their opposition to the reuse of their data for research purposes
* Vertebroplasties of more than one level
* History of spinal surgery or vertebroplasty near the level concerned

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient (≥18 years old) cared for at the HUS in interventional service for the realization of a vertebral cementoplasty of a single level
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-10-06 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Assess the interest of continuous visual monitoring of the fluoroscopy time by the operator on the dose delivered to the patient during an interventional radiology procedure performed under fluoroscopic control | up to 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Imagerie Interventionnelle - CHU de Strasbourg - France, Strasbourg, France